CLINICAL TRIAL: NCT01719003
Title: A 24-week Phase III Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Twice Daily Oral Administration of Empagliflozin + Metformin Compared With the Individual Components of Empagliflozin or Metformin in Drug Naive Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy Study of Empagliflozin and Metformin for 24 Weeks in Treatment Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1276.1; 2010-021375-92 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Metformin; BID protein, human; empagliflozin

ARMS (9):
- Empagliflozin low dose qd (Experimental): Empagliflozin low dose once daily
  Interventions: Drug: Empagliflozin low dose qd
- Empagliflozin high dose qd (Experimental): Empagliflozin high dose once daily
  Interventions: Drug: Empagliflozin high dose qd
- OL empa high dose + met 1000 mg bid (Experimental): Open label empagliflozin high dose split twice daily + metformin 1000 mg twice daily - Patients are no longer enrolled into this arm because of change in the inclusion criteria in protocol version 2.0 all patients are now enrolled into remaining double-blind arms. Patients already enrolled in the open-label arm according to protocol version 1.0 can complete the study.
  Interventions: Drug: Metformin 1000 mg bid; Drug: Empagliflozin high dose bid
- Empagliflozin low dose + met 500 mg bid (Experimental): Empagliflozin low dose split twice daily + metformin 500 mg twice daily
  Interventions: Drug: Metformin 500 mg bid; Drug: Empagliflozin low dose bid
- Empagliflozin low dose + met 1000 mg bid (Experimental): Empagliflozin low dose split twice daily + metformin 1000 mg twice daily
  Interventions: Drug: Empagliflozin low dose bid; Drug: Metformin 1000 mg bid
- Empagliflozin high dose + met 500 mg bid (Experimental): Empagliflozin high dose split twice daily + metformin 500 mg twice daily
  Interventions: Drug: Metformin 500 mg bid; Drug: Empagliflozin high dose bid
- Empagliflozin high dose + met 1000mg bid (Experimental): Empagliflozin high dose split twice daily + metformin 1000 mg twice daily
  Interventions: Drug: Metformin 1000 mg bid; Drug: Empagliflozin high dose bid
- Metformin 500 mg bid (Experimental): Metformin 500 mg twice daily
  Interventions: Drug: Metformin 500 mg bid
- Metformin 1000 mg bid (Experimental): Metformin 1000 mg twice daily
  Interventions: Drug: Metformin 1000 mg bid

INTERVENTIONS:
Drug: Metformin 500 mg bid — Metformin 500 mg twice daily
  Arms: Empagliflozin low dose + met 500 mg bid
Drug: Metformin 1000 mg bid — Metformin 1000 mg twice daily
  Arms: OL empa high dose + met 1000 mg bid
Drug: Empagliflozin low dose qd — Empagliflozin low dose once daily
  Arms: Empagliflozin low dose qd
Drug: Empagliflozin high dose qd — Empagliflozin high dose once daily
  Arms: Empagliflozin high dose qd
Drug: Empagliflozin low dose bid — Empagliflozin low dose split twice daily
  Arms: Empagliflozin low dose + met 500 mg bid
Drug: Metformin 500 mg bid — Metformin 500 mg twice daily
  Arms: Empagliflozin high dose + met 500 mg bid
Drug: Empagliflozin high dose bid — Empagliflozin high dose split twice daily
  Arms: OL empa high dose + met 1000 mg bid
Drug: Empagliflozin low dose bid — Empagliflozin low dose split twice daily
  Arms: Empagliflozin low dose + met 1000 mg bid
Drug: Metformin 1000 mg bid — Metformin 1000 mg twice daily
  Arms: Empagliflozin high dose + met 1000mg bid
Drug: Metformin 500 mg bid — Metformin 500 mg twice daily
  Arms: Metformin 500 mg bid
Drug: Metformin 1000 mg bid — Metformin 1000 mg twice daily
  Arms: Metformin 1000 mg bid
Drug: Empagliflozin high dose bid — Empagliflozin high dose split twice daily
  Arms: Empagliflozin high dose + met 1000mg bid
Drug: Metformin 1000 mg bid — Metformin 1000 mg twice daily
  Arms: Empagliflozin low dose + met 1000 mg bid
Drug: Empagliflozin high dose bid — Empagliflozin high dose split twice daily
  Arms: Empagliflozin high dose + met 500 mg bid

SUMMARY:
This study will investigate the efficacy and safety of two doses (high and low) of empagliflozin in combination with metformin (500 mg and 1000 mg) administered twice daily in patients with type 2 diabetes mellitus (T2DM). Study will compare four dose combinations of empagliflozin + metformin versus each individual component after 24 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent
2. Male and female patients on diet and exercise regimen who are drug-naive, defined as absence of any oral antidiabetic therapy for 12 weeks prior to randomization
3. HbA1c >=7.5% and <= 12% (>=58.5 mmol/mol and <=107.7 mmol/mol)
4. Body Mass Index (BMI) <= 45 kg/m2 at screening

Exclusion criteria:

1. Uncontrolled hyperglycemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second laboratory measurement (not on the same day)
2. Any antidiabetic drug within 12 weeks prior to randomization
3. Impaired renal function, defined as estimated creatinine clearance rate (eCCr) <60 ml/min (Cockcroft-Gault formula) as determined during screening and/or run-in period
4. Contraindications to metformin according to the local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1413 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (190):
- United States (41):
  - 1276.1.10014 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1276.1.10019 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1276.1.10044 Boehringer Ingelheim Investigational Site, Manley Hot Springs, Alaska
  - 1276.1.10010 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1276.1.10035 Boehringer Ingelheim Investigational Site, Searcy, Arkansas
  - 1276.1.10046 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1276.1.10006 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1276.1.10043 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1276.1.10009 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1276.1.10040 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1276.1.10045 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1276.1.10042 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1276.1.10001 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1276.1.10003 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1276.1.10026 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1276.1.10024 Boehringer Ingelheim Investigational Site, Oldsmar, Florida
  - 1276.1.10027 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1276.1.10023 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1276.1.10034 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1276.1.10032 Boehringer Ingelheim Investigational Site, Fall River, Massachusetts
  - 1276.1.10036 Boehringer Ingelheim Investigational Site, Bridgman, Michigan
  - 1276.1.10037 Boehringer Ingelheim Investigational Site, Hazelwood, Missouri
  - 1276.1.10007 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1276.1.10015 Boehringer Ingelheim Investigational Site, Union, New Jersey
  - 1276.1.10033 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1276.1.10022 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1276.1.10002 Boehringer Ingelheim Investigational Site, Lenoir, North Carolina
  - 1276.1.10005 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1276.1.10011 Boehringer Ingelheim Investigational Site, Gallipolis, Ohio
  - 1276.1.10030 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1276.1.10008 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1276.1.10013 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 1276.1.10017 Boehringer Ingelheim Investigational Site, Humboldt, Tennessee
  - 1276.1.10018 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.1.10025 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.1.10028 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.1.10016 Boehringer Ingelheim Investigational Site, Kingwood, Texas
  - 1276.1.10021 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1276.1.10041 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1276.1.10004 Boehringer Ingelheim Investigational Site, Manassas, Virginia
  - 1276.1.10012 Boehringer Ingelheim Investigational Site, Wenatchee, Washington
- Brazil (8):
  - 1276.1.55008 Boehringer Ingelheim Investigational Site, Belém
  - 1276.1.55003 Boehringer Ingelheim Investigational Site, Brasília
  - 1276.1.55006 Boehringer Ingelheim Investigational Site, Fortaleza
  - 1276.1.55007 Boehringer Ingelheim Investigational Site, Fortaleza
  - 1276.1.55009 Boehringer Ingelheim Investigational Site, Fortaleza
  - 1276.1.55004 Boehringer Ingelheim Investigational Site, Goiânia
  - 1276.1.55002 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1276.1.55001 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (11):
  - 1276.1.20003 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1276.1.20012 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1276.1.20008 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1276.1.20004 Boehringer Ingelheim Investigational Site, Antigonish, Nova Scotia
  - 1276.1.20005 Boehringer Ingelheim Investigational Site, Hawkesbury, Ontario
  - 1276.1.20013 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1276.1.20010 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1276.1.20006 Boehringer Ingelheim Investigational Site, Thornhill, Ontario
  - 1276.1.20007 Boehringer Ingelheim Investigational Site, Mirabel, Quebec
  - 1276.1.20002 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1276.1.20001 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Czechia (7):
  - 1276.1.42002 Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - 1276.1.42008 Boehringer Ingelheim Investigational Site, Olomouc
  - 1276.1.42007 Boehringer Ingelheim Investigational Site, Ostrava
  - 1276.1.42009 Boehringer Ingelheim Investigational Site, Pilsen
  - 1276.1.42003 Boehringer Ingelheim Investigational Site, Prague
  - 1276.1.42004 Boehringer Ingelheim Investigational Site, Prague
  - 1276.1.42010 Boehringer Ingelheim Investigational Site, Prague
- Egypt (4):
  - 1276.1.95001 Boehringer Ingelheim Investigational Site, Abbasia Cairo, Egypt
  - 1276.1.95003 Boehringer Ingelheim Investigational Site, Al Manial, Cairo, Egypt
  - 1276.1.95004 Boehringer Ingelheim Investigational Site, Alexandria
  - 1276.1.95002 Boehringer Ingelheim Investigational Site, El Darasa Cairo Egypt
- France (13):
  - 1276.1.33004 Boehringer Ingelheim Investigational Site, Behren-lès-Forbach
  - 1276.1.33012 Boehringer Ingelheim Investigational Site, Bersée
  - 1276.1.33005 Boehringer Ingelheim Investigational Site, Cournonterral
  - 1276.1.33007 Boehringer Ingelheim Investigational Site, Hautmont
  - 1276.1.33013 Boehringer Ingelheim Investigational Site, Paris
  - 1276.1.33001 Boehringer Ingelheim Investigational Site, Poitiers
  - 1276.1.33006 Boehringer Ingelheim Investigational Site, Saint-Génis-des-Fontaines
  - 1276.1.33003 Boehringer Ingelheim Investigational Site, Savonnières
  - 1276.1.33002 Boehringer Ingelheim Investigational Site, Thouars
  - 1276.1.33011 Boehringer Ingelheim Investigational Site, Thun-Saint-Amand
  - 1276.1.33010 Boehringer Ingelheim Investigational Site, Tours
  - 1276.1.33009 Boehringer Ingelheim Investigational Site, Vandome
  - 1276.1.33008 Boehringer Ingelheim Investigational Site, Vieux-Condé
- Germany (10):
  - 1276.1.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1276.1.49008 Boehringer Ingelheim Investigational Site, Celle
  - 1276.1.49006 Boehringer Ingelheim Investigational Site, Dortmund
  - 1276.1.49011 Boehringer Ingelheim Investigational Site, Dresden
  - 1276.1.49003 Boehringer Ingelheim Investigational Site, Essen
  - 1276.1.49007 Boehringer Ingelheim Investigational Site, Ingelheim
  - 1276.1.49014 Boehringer Ingelheim Investigational Site, Neuwied
  - 1276.1.49004 Boehringer Ingelheim Investigational Site, Offenbach
  - 1276.1.49002 Boehringer Ingelheim Investigational Site, Stuhr-Brinkum
  - 1276.1.49012 Boehringer Ingelheim Investigational Site, Teuchern
- Guatemala (5):
  - 1276.1.50002 Boehringer Ingelheim Investigational Site, Barbena Santa Rosa
  - 1276.1.50003 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1276.1.50005 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1276.1.50006 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1276.1.50001 Boehringer Ingelheim Investigational Site, Quetzaltenango
- Lebanon (4):
  - 1276.1.96001 Boehringer Ingelheim Investigational Site, Beirut
  - 1276.1.96002 Boehringer Ingelheim Investigational Site, El Chouf
  - 1276.1.96003 Boehringer Ingelheim Investigational Site, Saida
  - 1276.1.96004 Boehringer Ingelheim Investigational Site, Saida
- Malaysia (3):
  - 1276.1.60002 Boehringer Ingelheim Investigational Site, Ipoh, Perak
  - 1276.1.60001 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 1276.1.60003 Boehringer Ingelheim Investigational Site, Kubang Kerian
- Mexico (7):
  - 1276.1.52004 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1276.1.52007 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1276.1.52003 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1276.1.52002 Boehringer Ingelheim Investigational Site, Mexico City
  - 1276.1.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1276.1.52006 Boehringer Ingelheim Investigational Site, San Lucas Tepetlcalco
  - 1276.1.52005 Boehringer Ingelheim Investigational Site, Zapopan
- Peru (5):
  - 1276.1.51001 Boehringer Ingelheim Investigational Site, Lima
  - 1276.1.51002 Boehringer Ingelheim Investigational Site, Lima
  - 1276.1.51003 Boehringer Ingelheim Investigational Site, Lima
  - 1276.1.51004 Boehringer Ingelheim Investigational Site, Lima
  - 1276.1.51005 Boehringer Ingelheim Investigational Site, Lima
- Philippines (9):
  - 1276.1.63009 Boehringer Ingelheim Investigational Site, Cebu City, Cebu
  - 1276.1.63002 Boehringer Ingelheim Investigational Site, Cebu City, Philippines
  - 1276.1.63004 Boehringer Ingelheim Investigational Site, Davao City
  - 1276.1.63003 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1276.1.63006 Boehringer Ingelheim Investigational Site, Manila
  - 1276.1.63001 Boehringer Ingelheim Investigational Site, Marikina City
  - 1276.1.63005 Boehringer Ingelheim Investigational Site, Maybunga, Pasig City
  - 1276.1.63007 Boehringer Ingelheim Investigational Site, San Juan City
  - 1276.1.63008 Boehringer Ingelheim Investigational Site, Tarlac City
- Russia (12):
  - 1276.1.70012 Boehringer Ingelheim Investigational Site, Barnaul
  - 1276.1.70011 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1276.1.70015 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1276.1.70016 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1276.1.70018 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1276.1.70007 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 1276.1.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1276.1.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1276.1.70017 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1276.1.70009 Boehringer Ingelheim Investigational Site, Saratov
  - 1276.1.70010 Boehringer Ingelheim Investigational Site, Smolensk
  - 1276.1.70013 Boehringer Ingelheim Investigational Site, Yaroslavl
- Serbia (8):
  - 1276.1.38104 Boehringer Ingelheim Investigational Site, Belgrade
  - 1276.1.38105 Boehringer Ingelheim Investigational Site, Belgrade
  - 1276.1.38106 Boehringer Ingelheim Investigational Site, Belgrade
  - 1276.1.38107 Boehringer Ingelheim Investigational Site, Belgrade
  - 1276.1.38103 Boehringer Ingelheim Investigational Site, Kragujevac
  - 1276.1.38101 Boehringer Ingelheim Investigational Site, Niš
  - 1276.1.38108 Boehringer Ingelheim Investigational Site, Novi Sad
  - 1276.1.38102 Boehringer Ingelheim Investigational Site, Zaječar
- South Korea (10):
  - 1276.1.82006 Boehringer Ingelheim Investigational Site, Deagu
  - 1276.1.82010 Boehringer Ingelheim Investigational Site, Goyang
  - 1276.1.82001 Boehringer Ingelheim Investigational Site, Incheon
  - 1276.1.82009 Boehringer Ingelheim Investigational Site, Pusan
  - 1276.1.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1276.1.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1276.1.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1276.1.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1276.1.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1276.1.82003 Boehringer Ingelheim Investigational Site, Wŏnju
- Spain (8):
  - 1276.1.34048 Boehringer Ingelheim Investigational Site, Alicante
  - 1276.1.34050 Boehringer Ingelheim Investigational Site, Alzira
  - 1276.1.34028 Boehringer Ingelheim Investigational Site, Madrid
  - 1276.1.34045 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 1276.1.34034 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1276.1.34027 Boehringer Ingelheim Investigational Site, Salamanca
  - 1276.1.34052 Boehringer Ingelheim Investigational Site, Tarragona
  - 1276.1.34051 Boehringer Ingelheim Investigational Site, Zaragoza
- Taiwan (6):
  - 1276.1.88005 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1276.1.88002 Boehringer Ingelheim Investigational Site, New Taipei City
  - 1276.1.88001 Boehringer Ingelheim Investigational Site, Taichung
  - 1276.1.88003 Boehringer Ingelheim Investigational Site, Taichung
  - 1276.1.88004 Boehringer Ingelheim Investigational Site, Taichung
  - 1276.1.88006 Boehringer Ingelheim Investigational Site, Taipei
- Thailand (3):
  - 1276.1.66001 Boehringer Ingelheim Investigational Site, Bangkok, Thailand
  - 1276.1.66003 Boehringer Ingelheim Investigational Site, Bangkok, Thailand
  - 1276.1.66002 Boehringer Ingelheim Investigational Site, Nakhon Ratchasima
- Turkey (Türkiye) (6):
  - 1276.1.90003 Boehringer Ingelheim Investigational Site, Ankara
  - 1276.1.90004 Boehringer Ingelheim Investigational Site, Antalya
  - 1276.1.90006 Boehringer Ingelheim Investigational Site, Denizli
  - 1276.1.90002 Boehringer Ingelheim Investigational Site, Erzurum
  - 1276.1.90005 Boehringer Ingelheim Investigational Site, Istanbul
  - 1276.1.90001 Boehringer Ingelheim Investigational Site, Izmir
- United Kingdom (10):
  - 1276.1.44002 Boehringer Ingelheim Investigational Site, Bolton
  - 1276.1.44001 Boehringer Ingelheim Investigational Site, Bradford-on-Avon
  - 1276.1.44005 Boehringer Ingelheim Investigational Site, Chippenham
  - 1276.1.44006 Boehringer Ingelheim Investigational Site, Dagenham
  - 1276.1.44004 Boehringer Ingelheim Investigational Site, Doncaster
  - 1276.1.44008 Boehringer Ingelheim Investigational Site, Glasgow
  - 1276.1.44003 Boehringer Ingelheim Investigational Site, Leeds
  - 1276.1.44007 Boehringer Ingelheim Investigational Site, Manchester
  - 1276.1.44011 Boehringer Ingelheim Investigational Site, Mortimer
  - 1276.1.44009 Boehringer Ingelheim Investigational Site, Sandbach

REFERENCES:
- [Derived] Hadjadj S, Rosenstock J, Meinicke T, Woerle HJ, Broedl UC. Initial Combination of Empagliflozin and Metformin in Patients With Type 2 Diabetes. Diabetes Care. 2016 Oct;39(10):1718-28. doi: 10.2337/dc16-0522. Epub 2016 Aug 4. PMID 27493136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With the first global protocol amendment (13-Dec-2012), the HbA1c inclusion criterion changed and further enrolment in the open label (OL) group was stopped, but the patients already entered in the OL group could continue until the scheduled end of the study.
Pre-assignment Details: Patients with an (Glycosylated Haemoglobin) HbA1c >10.0% at screening and meeting all other inclusion criteria were initially directly included in an OL treatment group
Groups:
- Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid: Oral administration of Empagliflozin 12.5 mg and Metformin 1000 mg twice daily (bid)
- Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid: Oral administration of Empagliflozin 12.5 mg and Metformin 500 mg bid
- Empagliflozin 5 mg Bid + Metformin 1000 mg Bid: Oral administration of Empagliflozin 5 mg and Metformin 1000 mg bid
- Empagliflozin 5 mg Bid + Metformin 500 mg Bid: Oral administration of Empagliflozin 5 mg and Metformin 500 mg bid
- Empagliflozin 25 mg qd: Oral administration of Empagliflozin 25 mg once daily (qd)
- Empagliflozin 10 mg qd: Oral administration of Empagliflozin 10 mg qd
- Metformin 1000 mg Bid: Oral administration of Metformin 1000 mg bid
- Metformin 500 mg Bid: Oral administration of Metformin 500 mg bid
- Empagliflozin 12.5 mg Bid + Metformin 1000 mg Bid OL: Oral administration of Empagliflozin 12.5 mg and Metformin 1000 mg bid in an open label (OL)
Period: Overall Study
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid | Empagliflozin 12.5 mg Bid + Metformin 1000 mg Bid OL
Started | 170 | 170 | 171 | 169 | 167 | 172 | 170 | 171 | 53
Completed | 161 | 153 | 154 | 156 | 150 | 160 | 150 | 151 | 49
Not Completed | 9 | 17 | 17 | 13 | 17 | 12 | 20 | 20 | 4
Not completed — Non compliant with protocol | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 0
Not completed — Adverse Event | 6 | 5 | 4 | 3 | 4 | 3 | 6 | 5 | 0
Not completed — Lost to Follow-up | 0 | 6 | 7 | 2 | 3 | 4 | 3 | 2 | 2
Not completed — Refusal to continue, not due to AE | 2 | 5 | 4 | 4 | 4 | 3 | 8 | 7 | 1
Not completed — Reason other than those specified | 0 | 0 | 2 | 3 | 4 | 1 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): FAS comprised all randomised patients treated with at least 1 dose of trial medication, with a baseline and at least 1 on-treatment HbA1c assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid | Total
Number analyzed (Participants) | 169 | 165 | 167 | 161 | 164 | 169 | 164 | 168 | 1327
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (10.7) | 51.0 (10.7) | 52.3 (11.3) | 52.2 (11.7) | 53.3 (10.7) | 53.1 (10.7) | 51.6 (10.8) | 53.4 (10.9) | 52.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 60 | 68 | 64 | 81 | 72 | 72 | 82 | 580
  Male | 88 | 105 | 99 | 97 | 83 | 97 | 92 | 86 | 747

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin) Change From Baseline at Week 24
Description: Change from baseline in HbA1c (%) after 24 weeks of treatment. "Baseline" refers to the last observation before the start of any randomised trial treatment medication. Means presented are the adjusted means
Time Frame: baseline and 24 weeks
Population: FAS observed cases (OC) (Only patients with available data are analysed)
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid
Number analyzed (Participants) | 159 | 149 | 151 | 153 | 143 | 156 | 146 | 142
percentage of HbA1c | -2.08 (0.08) | -1.93 (0.08) | -2.07 (0.08) | -1.98 (0.08) | -1.36 (0.08) | -1.35 (0.08) | -1.75 (0.09) | -1.18 (0.08)
Statistical Analysis 1: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid vs Metformin 1000 mg Bid; Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach comparing the change from baseline of HbA1c (in units of %) after 24 weeks of double-blind treatment; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; 'Baseline HbA1c':linear covariate;'treatment','baseline renal function','region','visit' & 'visit by treatment interaction':fixed effects; Adjusted mean = -0.33, 95% CI 2-sided [-0.56 to -0.10], Standard Error of Mean 0.12 — Empagliflozin 12.5 mg bid+ Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 2: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid vs Empagliflozin 25 mg qd; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -0.72, 95% CI 2-sided [-0.95 to -0.48], Standard Error of Mean 0.12 — Empagliflozin 12.5 mg bid+ Metformin 1000 mg bid minus Empagliflozin 25 mg qd
Statistical Analysis 3: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -0.75, 95% CI 2-sided [-0.98 to -0.51], Standard Error of Mean 0.12 — Empagliflozin 12.5 mg bid+ Metformin 500 mg bid minus Metformin 500 mg bid
Statistical Analysis 4: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid vs Empagliflozin 25 mg qd; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -0.57, 95% CI 2-sided [-0.81 to -0.34], Standard Error of Mean 0.12 — Empagliflozin 12.5 mg bid+ Metformin 500 mg bid minus Empagliflozin 25 mg qd
Statistical Analysis 5: Comparison: Empagliflozin 5 mg Bid + Metformin 1000 mg Bid vs Metformin 1000 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -0.33, 95% CI 2-sided [-0.56 to -0.09], Standard Error of Mean 0.12 — Empagliflozin 5 mg bid + Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 6: Comparison: Empagliflozin 5 mg Bid + Metformin 1000 mg Bid vs Empagliflozin 10 mg qd; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -0.72, 95% CI 2-sided [-0.95 to -0.49], Standard Error of Mean 0.12 — Empagliflozin 5 mg bid + Metformin 1000 mg bid minus Empagliflozin 10 mg qd
Statistical Analysis 7: Comparison: Empagliflozin 5 mg Bid + Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -0.79, 95% CI 2-sided [-1.03 to -0.56], Standard Error of Mean 0.12 — Empagliflozin 5 mg bid + Metformin 500 mg bid minus Metformin 500 mg bid
Statistical Analysis 8: Comparison: Empagliflozin 5 mg Bid + Metformin 500 mg Bid vs Empagliflozin 10 mg qd; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -0.63, 95% CI 2-sided [-0.86 to -0.40], Standard Error of Mean 0.12 — Empagliflozin 5 mg bid + Metformin 500 mg bid minus Empagliflozin 10 mg qd
Statistical Analysis 9: Comparison: Empagliflozin 25 mg qd vs Metformin 1000 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The noninferiority of empagliflozin 10 mg qd against metformin 1000 mg bid were to be tested for HbA1c change from baseline to Week 24 at the level of α=0.025 (one-sided), through application of a non-inferiority margin of 0.35%; p = 0.6246, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = 0.39, 95% CI 2-sided [0.15 to 0.62], Standard Error of Mean 0.12 — Empagliflozin 25 mg qd minus Metformin 1000 mg bid
Statistical Analysis 10: Comparison: Empagliflozin 10 mg qd vs Metformin 1000 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 9]; p = 0.6558, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean = 0.40, 95% CI 2-sided [0.16 to 0.63], Standard Error of Mean 0.12 — Empagliflozin 10 mg qd minus Metformin 1000 mg bid

2. Secondary Outcome: FPG (Fasting Plasma Glucose) Change From Baseline at Week 24
Description: Change from baseline in FPG (mg/dL) after 24 weeks of treatment. "Baseline" refers to the last observation before the start of any randomised trial treatment medication. Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS observed cases (OC) (Only patients with available data are analysed)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid
Number analyzed (Participants) | 158 | 146 | 146 | 153 | 139 | 154 | 145 | 139
mg/dL | -51.0 (2.4) | -44.0 (2.4) | -47.8 (2.4) | -45.5 (2.4) | -28.0 (2.5) | -32.9 (2.4) | -32.1 (2.4) | -17.2 (2.5)
Statistical Analysis 1: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid vs Metformin 1000 mg Bid; Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach comparing the change from baseline of FPG after 24 weeks of double-blind treatment; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Since previous step in the hierarchical testing failed (primary measure analyses 9 and 10), the analyses for secondary measures of FPG and body weight are considered exploratory and not confirmatory; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -18.8, 95% CI 2-sided [-25.5 to -12.2], Standard Error of Mean 3.4 — Empagliflozin 12.5 mg bid+ Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 2: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid vs Empagliflozin 25 mg qd; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -23.0, 95% CI 2-sided [-29.7 to -16.3], Standard Error of Mean 3.4 — Empagliflozin 12.5 mg bid+ Metformin 1000 mg bid minus Empagliflozin 25 mg qd
Statistical Analysis 3: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -26.7, 95% CI 2-sided [-33.5 to -20.0], Standard Error of Mean 3.4 — Empagliflozin 12.5 mg bid+ Metformin 500 mg bid minus Metformin 500 mg bid
Statistical Analysis 4: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid vs Empagliflozin 25 mg qd; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -16.0, 95% CI 2-sided [-22.8 to -9.2], Standard Error of Mean 3.4 — Empagliflozin 12.5 mg bid+ Metformin 500 mg bid minus Empagliflozin 25 mg qd
Statistical Analysis 5: Comparison: Empagliflozin 5 mg Bid + Metformin 1000 mg Bid vs Metformin 1000 mg Bid; Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach comparing the change from baseline of FPG of double-blind treatment; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -15.6, 95% CI 2-sided [-22.3 to -8.9], Standard Error of Mean 3.4 — Empagliflozin 5 mg bid + Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 6: Comparison: Empagliflozin 5 mg Bid + Metformin 1000 mg Bid vs Empagliflozin 10 mg qd; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -14.8, 95% CI 2-sided [-21.4 to -8.2], Standard Error of Mean 3.4 — Empagliflozin 5 mg bid + Metformin 1000 mg bid minus Empagliflozin 10 mg qd
Statistical Analysis 7: Comparison: Empagliflozin 5 mg Bid + Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -28.2, 95% CI 2-sided [-35.0 to -21.5], Standard Error of Mean 3.4 — Empagliflozin 5 mg bid + Metformin 500 mg bid minus Metformin 500 mg bid
Statistical Analysis 8: Comparison: Empagliflozin 5 mg Bid + Metformin 500 mg Bid vs Empagliflozin 10 mg qd; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -12.6, 95% CI 2-sided [-19.1 to -6.0], Standard Error of Mean 3.4 — Empagliflozin 5 mg bid + Metformin 500 mg bid minus Empagliflozin 10 mg qd

3. Secondary Outcome: Body Weight Change From Baseline at Week 24
Description: Change from baseline in body weight (kg) after 24 weeks of treatment. "Baseline" refers to the last observation before the start of any randomised trial treatment. medication. Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS observed cases (OC) (Only patients with available data are analysed)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid
Number analyzed (Participants) | 160 | 149 | 150 | 155 | 143 | 155 | 148 | 140
kg | -3.78 (0.29) | -3.04 (0.30) | -3.48 (0.30) | -2.77 (0.30) | -2.38 (0.30) | -2.39 (0.29) | -1.27 (0.30) | -0.52 (0.30)
Statistical Analysis 1: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid vs Metformin 1000 mg Bid; Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach comparing the change from baseline of body weight after 24 weeks of double-blind treatment; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -2.50, 95% CI 2-sided [-3.33 to -1.68], Standard Error of Mean 0.42 — Empagliflozin 12.5 mg bid+ Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 2: Comparison: Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -2.52, 95% CI 2-sided [-3.35 to -1.69], Standard Error of Mean 0.42 — Empagliflozin 12.5 mg bid+ Metformin 500 mg bid minus Metformin 500 mg bid
Statistical Analysis 3: Comparison: Empagliflozin 5 mg Bid + Metformin 1000 mg Bid vs Metformin 1000 mg Bid; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean = -2.20, 95% CI 2-sided [-3.03 to -1.37], Standard Error of Mean 0.42 — Empagliflozin 5 mg bid + Metformin 1000 mg bid minus Metformin 1000 mg bid
Statistical Analysis 4: Comparison: Empagliflozin 5 mg Bid + Metformin 500 mg Bid vs Metformin 500 mg Bid; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean = -2.26, 95% CI 2-sided [-3.09 to -1.43], Standard Error of Mean 0.42 — Empagliflozin 5 mg bid + Metformin 500 mg bid minus Metformin 500 mg bid

ADVERSE EVENTS:
Time Frame: Adverse events with an onset after the first dose of randomised trial medication up to a period of 7 days after the last dose (Up to 237 days)
Arm/Group | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid | Empagliflozin 5 mg Bid + Metformin 500 mg Bid | Empagliflozin 25 mg qd | Empagliflozin 10 mg qd | Metformin 1000 mg Bid | Metformin 500 mg Bid | Empagliflozin 12.5 mg Bid + Metformin 1000 mg Bid OL
Serious Adverse Events (participants affected / at risk) | 2/170 | 6/170 | 3/171 | 2/169 | 3/167 | 1/172 | 3/170 | 3/171 | 2/53
Other Adverse Events (participants affected / at risk) | 48/170 | 40/170 | 35/171 | 42/169 | 41/167 | 36/172 | 53/170 | 38/171 | 16/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid (N=170) | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid (N=170) | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid (N=171) | Empagliflozin 5 mg Bid + Metformin 500 mg Bid (N=169) | Empagliflozin 25 mg qd (N=167) | Empagliflozin 10 mg qd (N=172) | Metformin 1000 mg Bid (N=170) | Metformin 500 mg Bid (N=171) | Empagliflozin 12.5 mg Bid + Metformin 1000 mg Bid OL (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 12.5 mg Bid+ Metformin 1000 mg Bid (N=170) | Empagliflozin 12.5 mg Bid+ Metformin 500 mg Bid (N=170) | Empagliflozin 5 mg Bid + Metformin 1000 mg Bid (N=171) | Empagliflozin 5 mg Bid + Metformin 500 mg Bid (N=169) | Empagliflozin 25 mg qd (N=167) | Empagliflozin 10 mg qd (N=172) | Metformin 1000 mg Bid (N=170) | Metformin 500 mg Bid (N=171) | Empagliflozin 12.5 mg Bid + Metformin 1000 mg Bid OL (N=53)
Diarrhoea (Gastrointestinal disorders) | 12 | 6 | 5 | 9 | 6 | 2 | 24 | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 8 | 4 | 7 | 5 | 5 | 10 | 3
Urinary tract infection (Infections and infestations) | 18 | 17 | 12 | 9 | 13 | 12 | 14 | 12 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 6 | 8 | 15 | 11 | 15 | 8 | 7 | 2
Dizziness (Nervous system disorders) | 6 | 9 | 4 | 5 | 3 | 4 | 4 | 7 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 4 | 2 | 3
Nausea (Gastrointestinal disorders) | 6 | 4 | 5 | 5 | 1 | 1 | 3 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 1 | 0 | 1 | 2 | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights